CLINICAL TRIAL: NCT01232751
Title: The Effect of Isoflavone Supplement Intake on Gene-expression in Postmenopausal Women
Brief Title: Effects of Isoflavones on Gene-expression
Acronym: ISO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Principal Investigator, Lisette de Groot, (Vera van der Velpen), Wageningen University
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: NL 32375.081.10
Record Dates: First submitted 2010-10-21; First posted 2010-11-02 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Postmenopause
Keywords: health; women

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Isoflavone supplement — The participants will consume 2 times 2 supplements per day, which will lead to a daily dose of 114 mg. (HPLC analysis confirmed an aglycone isoflavone content of 28.41 mg per supplement)
  Other Names: Phytosoya forte (35mg) from the company Arkopharma

SUMMARY:
Alleged benefits experienced by the consumption of soy in Asian countries have been attributed to the isoflavone content of soy products. Amongst other benefits, isoflavones are believed to relieve menopausal symptoms and are therefore often consumed in supplement form in Western countries. These supplements contain relatively high amounts of isoflavones, and the question is if these concentrations still exert beneficial effects or whether negative effects become dominant. Therefore, the investigators will study the effect of intake of one dose of isoflavones, as compared to placebo, for eight weeks on gene-expression in Peripheral Blood Mononuclear Cells (PBMCs) in post-menopausal, equol-producing women.

DETAILED DESCRIPTION:
Primary Objective: to determine the effect of intake of one dose of isoflavones, as compared to placebo, for eight weeks on gene-expression in Peripheral Blood Mononuclear Cells (PBMCs) in post-menopausal, equol-producing women.

Secondary Objectives: to determine the association between isoflavone plasma levels and gene-expression in PBMCs; to determine the variation of isoflavone plasma levels between subjects after intake of isoflavones for four and eight weeks; to explore whether PBMC gene-expression markers identified after 8 weeks isoflavone intervention are already present after 4 weeks intervention; to explore whether the severity of previous menopausal complaints is related to the effect of isoflavones on PBMC gene-expression; and to explore the association between isoflavone levels in plasma and spot urine.

Study design: Double-blind placebo controlled crossover intervention study

Study population: Thirty-six healthy females, 45-70 years, post-menopausal and equol-producing

Intervention: Two intervention periods of eight weeks with a isoflavone supplement or a placebo and a washout period of 8 weeks in between.

Main study parameters/endpoints: The main study parameter is gene-expression in PBMCs measured by micro-arrays.

ELIGIBILITY:
Inclusion Criteria:

* 45-70 years
* Equol producer
* Post-menopausal (Follicle Stimulating Hormone (FSH) >40 UI/L) or
* menstrual cycle absent for more than 1 year.

Exclusion Criteria:

* current use of contraceptives containing hormones
* current use of hormone replacement therapy
* regular soy product use (more than once a week)
* regular isoflavone supplement use (more than once a week)
* current use of medication containing sex hormones or sex hormone-triggering compounds
* current use of anti-inflammatory medicines
* use of antibiotics in the past 6 months
* severe heart disease
* thyroid disorders
* removed thyroid gland
* complete ovariectomy
* prior diagnosis of cancer in medical history
* alcohol and drug abuse
* current smoker
* Body Mass Index (BMI) >35 kg/m2
* allergy to soy (products)

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Gene-expression measured by micro-arrays | gene-expression after 8 weeks of exposure to the isoflavone supplement
  Gene expression changes will be assessed in PBMCs using whole genome Affymetrix microarrays. The gene expression changes after exposure to the isoflavone supplement will be compared to the changes after exposure to the placebo.
Gene-expression measured by micro-arrays | after 8 weeks of exposure to the placebo
  Gene expression changes will be assessed in PBMCs using whole genome Affymetrix microarrays. The gene expression changes after exposure to the isoflavone supplement will be compared to the changes after exposure to the placebo.

SECONDARY OUTCOMES:
Isoflavone levels in plasma and spoturine | after 0 weeks of exposure to the isoflavone supplement
  levels of the isoflavones genistein, dihydrogenistein, daidzein, dihydrodaidzein, equol and glycitein will be measured with High performance liquid chromatography (HPLC). Following the intention to treat analysis, these concentration markers will be determined in order to correlate the gene-expression measured with quantitative real-time polymerase chain reaction (QPCR) with the isoflavone plasma levels, and to stratify for the plasma levels in per protocol analysis.
Isoflavone levels in plasma and spoturine | after 4 weeks of exposure to the isoflavone supplement
  levels of the isoflavones genistein, dihydrogenistein, daidzein, dihydrodaidzein, equol and glycitein will be measured with HPLC. Following the intention to treat analysis, these concentration markers will be determined in order to correlate the gene-expression measured with QPCR with the isoflavone plasma levels, and to stratify for the plasma levels in per protocol analysis.
Isoflavone levels in plasma and spoturine | after 8 weeks of exposure to the isoflavone supplement
  levels of the isoflavones genistein, dihydrogenistein, daidzein, dihydrodaidzein, equol and glycitein will be measured with HPLC. Following the intention to treat analysis, these concentration markers will be determined in order to correlate the gene-expression measured with QPCR with the isoflavone plasma levels, and to stratify for the plasma levels in per protocol analysis.
Isoflavone levels in plasma and spoturine | after 0 weeks of exposure to the placebo
  levels of the isoflavones genistein, dihydrogenistein, daidzein, dihydrodaidzein, equol and glycitein will be measured with HPLC. Following the intention to treat analysis, these concentration markers will be determined in order to correlate the gene-expression measured with QPCR with the isoflavone plasma levels, and to stratify for the plasma levels in per protocol analysis.
Isoflavone levels in plasma and spoturine | after 4 weeks of exposure to the placebo
  levels of the isoflavones genistein, dihydrogenistein, daidzein, dihydrodaidzein, equol and glycitein will be measured with HPLC. Following the intention to treat analysis, these concentration markers will be determined in order to correlate the gene-expression measured with QPCR with the isoflavone plasma levels, and to stratify for the plasma levels in per protocol analysis.
Isoflavone levels in plasma and spoturine | after 8 weeks of exposure to the placebo
  levels of the isoflavones genistein, dihydrogenistein, daidzein, dihydrodaidzein, equol and glycitein will be measured with HPLC. Following the intention to treat analysis, these concentration markers will be determined in order to correlate the gene-expression measured with QPCR with the isoflavone plasma levels, and to stratify for the plasma levels in per protocol analysis.
Confirmation of gene-expression with quantitative real time polymerase chain reaction (QPCR) | after 0 weeks of exposure to the isoflavone supplement
  Ten genes per sample will be verified with QPCR. PBMCs from the subjects are available at time points before, halfway and after the two intervention periods. On the basis of the micro-array results it will be decided which genes from which samples will be quantified.
Confirmation of gene-expression with quantitative real time polymerase chain reaction (QPCR) | after 4 weeks of exposure to the isoflavone supplement
  Ten genes per sample will be verified with QPCR. PBMCs from the subjects are available at time points before, halfway and after the two intervention periods. On the basis of the micro-array results it will be decided which genes from which samples will be quantified.
Confirmation of gene-expression with quantitative real time polymerase chain reaction (QPCR) | after 0 weeks of exposure to the placebo
  Ten genes per sample will be verified with QPCR. PBMCs from the subjects are available at time points before, halfway and after the two intervention periods. On the basis of the micro-array results it will be decided which genes from which samples will be quantified.
Confirmation of gene-expression with quantitative real time polymerase chain reaction (QPCR) | after 8 weeks of exposure to the isoflavone supplement
  Ten genes per sample will be verified with QPCR. PBMCs from the subjects are available at time points before, halfway and after the two intervention periods. On the basis of the micro-array results it will be decided which genes from which samples will be quantified.
Confirmation of gene-expression with quantitative real time polymerase chain reaction (QPCR) | after 4 weeks of exposure to the placebo
  Ten genes per sample will be verified with QPCR. PBMCs from the subjects are available at time points before, halfway and after the two intervention periods. On the basis of the micro-array results it will be decided which genes from which samples will be quantified.
Confirmation of gene-expression with quantitative real time polymerase chain reaction (QPCR) | after 8 weeks of exposure to the placebo
  Ten genes per sample will be verified with QPCR. PBMCs from the subjects are available at time points before, halfway and after the two intervention periods. On the basis of the micro-array results it will be decided which genes from which samples will be quantified.

CONTACTS AND LOCATIONS:
Overall Officials: Pieter van 't Veer, Professor, Principal Investigator — Wageningen University
Locations (1):
- Wageningen University, Wageningen, Gelderland, Netherlands

REFERENCES:
- [Derived] van der Velpen V, Geelen A, Schouten EG, Hollman PC, Afman LA, van 't Veer P. Estrogen receptor-mediated effects of isoflavone supplementation were not observed in whole-genome gene expression profiles of peripheral blood mononuclear cells in postmenopausal, equol-producing women. J Nutr. 2013 Jun;143(6):774-80. doi: 10.3945/jn.113.174037. Epub 2013 Apr 24. PMID 23616509